CLINICAL TRIAL: NCT05172206
Title: Symptom-based Rehabilitation Compared to Usual Care in Post-COVID - a Randomized Controlled Trial
Acronym: RELOAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: Bavarian State Office for Health and Food Safety (Unknown); Praxis im Zentrum Erlangen (Unknown); Pneumologen Lichterfelde Berlin (Unknown); Pneumopraxis Marburg (Unknown); COVID ambulance Philipps-University Marburg (Unknown); Pneumologie Elisenhof Munich (Unknown); COVID ambulance Pneumology LMU Munich (Unknown); COVID ambulance psychology LMU Munich (Unknown); University Clinic Augsburg (Unknown); COVID ambulance Schön Klinik Schönau (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Rembert Koczulla, Professor, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RELOAD
Record Dates: First submitted 2021-12-22; First posted 2021-12-29 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: COVID-19; Long-COVID
Keywords: rehabilitation; intervention; quality of life; long-COVID; post-COVID syndrome; sequelae; recovery
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Symptom-focused Rehabilitation (Active Comparator): Patients in this arm will be referred to a 3-week inpatient comprehensive rehabilitation program. Initially, patients will be classified into one out of three clusters namely: Cluster A (Fatigue), Cluster B (cognition), or Cluster C (physical). The content of the rehabilitation program will be individually adapted according to the patient's most relevant symptom cluster.
  Interventions: Other: symptom-focused rehabilitation
- Usual Care (Other): Patients in this arm do not receive any intervention beyond usual care during the study phase. However, all patients in this group will get the opportunity to also receive a rehabilitation program after the study phase.
  Interventions: Other: usual care

INTERVENTIONS:
Other: symptom-focused rehabilitation — Patients in this arm will be referred to a 3-week inpatient comprehensive rehabilitation program. Initially, patients will be classified into one out of three clusters namely: Cluster A (Fatigue), Cluster B (cognition), or Cluster C (physical). The content of the rehabilitation program will be individually adapted according to the patient's most relevant symptom cluster.
  Arms: Symptom-focused Rehabilitation
Other: usual care — Patients in this arm do not receive any intervention beyond usual care during the study phase. However, all patients in this group will get the opportunity to also receive a rehabilitation program after the study phase.
  Arms: Usual Care

SUMMARY:
Inpatient, multimodal rehabilitation represents one of the most important interventions in the disease management of post/long COVID. Different professional societies, including the German Society of Pneumology and the European Respiratory Society, recommend rehabilitation intervention to reduce the sequelae of COVID-19. However, from the perspective of science and practice, there are relevant areas that have been insufficiently investigated and are essential for the treatment success of post/long COVID patients:

* Differentiation of rehabilitation effects from natural recovery after COVID-19.
* Lack of personalized and symptom-based treatment approaches that can address the heterogeneity of symptoms in post/long COVID
* Lack of uniform, high-quality rehabilitation standards in post-/long-COVID.

Therefore, post-COVID patients will be recruited at several post-COVID practices around Germany and randomized to receive (A) a rehabilitation program or (B) usual care. The primary objective of this randomized controlled trial (RCT) is to investigate whether a 3-week symptom-oriented, inpatient, multidisciplinary rehabilitation intervention, whose content focus is standardized according to cluster assignment (fatigue, cognition, soma), has a positive effect on the quality of life (primary outcome) in post-COVID syndrome patients compared to a usual care group (standard outpatient care). All study participants will be provided with a continuous telemonitoring system (SaniQ app) throughout the study period. After the interventional phase, there will be a 3 months follow-up assessment to evaluate the maintenance effects of COVID rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Post-COVID Syndrome according to World Health Organisation definition (persistent symptoms for at least 3 months after PCR-test confirmed SARS-CoV 2 infection)

Exclusion Criteria:

* no walking ability
* not able to operate smartphone apps
* rehabilitation program within the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Change from baseline Quality of life assessed by Short Form - 12 Questionnaire at week 4 and week 12 | baseline, week 4, week 12
  the scale of the physical and mental Health component summary score ranges from minimum 0 to maximum 100 points with higher scores indicating better quality of life

SECONDARY OUTCOMES:
Change from baseline COVID-related symptoms at week 4 and week 12 | baseline, week 4, week 12
  the number of COVID-symptoms will recorded as well as their intensity will be rated on a scale from 0 [not relevant] until 10 [very severe symptom].
Change from baseline lung function at week 4 and week 12 | baseline, week 4, week 12
  following Parameters will be collected: forced expiratory volume in 1 sec, peak flow, forced vital capacity, total lung capacity, diffusion lung capacity for carbonmonoxide
Change from baseline blood gas analysis at week 4 and week 12 | baseline, week 4, week 12
  following parameters will be collected at rest and at the end of an incremental cycle test: partial pressure for oxygen and carbon dioxide
Change from baseline Cardiac Doppler echocardiography at week 4 and week 12 | baseline, week 4, week 12
  Left and right heart echocardiography will be performed
Change from baseline laboratory parameters at week 4 and week 12 | baseline, week 4, week 12
  blood samples will be taken from venous blood
Change from baseline exercise performance at week 4 and week 12 | baseline, week 4, week 12
  incremental cardiopulmonary exercise testing will be performed with spirometry
Change from baseline health care service needs at week 4 and week 12 | baseline, week 4, week 12
  Number of visits at the general practitioner, pulmonologist, psychologist, physiotherapist, COVID-ambulance, hospital admission until the last visit will be recorded
Change from baseline working capability at week 4 and week 12 | baseline, week 4, week 12
  number of days of incapacity to work until the last visit will be recorded
Change from baseline sleep quality at week 4 and week 12 | baseline, week 4, week 12
  Sleep quality will be assessed by using the Pittsburgh Sleep Quality Index (total score ranges from 0 to 21 with higher scores indicating higher impairment)
Change from baseline sleep quality at week 4 and week 12 | baseline, week 4, week 12
  daytime sleepiness will be assessed by using the Epworth Sleepiness Scale (total score ranges from 0 to 24 with higher scores indicating higher impairment)
Change from baseline Depression status assessed by Patient Health Questionnaire 9 | baseline, week 4, week 12
  the total score ranges from 0 to 27 points with higher scores indicating worse Depression symptoms
Change from baseline Anxiety status assessed by Generalized Anxiety Disorder Scale 7 | baseline, week 4, week 12
  the total score ranges from 0 to 21 points with higher scores indicating more anxiety symptoms
Change from baseline resilience assessed by resilience scale 13 | baseline, week 4, week 12
  the total score ranges from 13 to 91 points with higher scores indicating higher resilience
Change from baseline cognitive status assessed by Montreal Cognitive Assessment Test | baseline, week 4, week 12
  the total score ranges from 0 to 30 points with higher scores indicating a better cognitive status
Change from baseline dyspnea assessed by Modified Medical Research Counsil score at week 4 and week 12 | baseline, week 4, week 12
  the total score ranges from 0 to 4 points with higher scores indicating more dyspnea
Change from baseline dysfunctional breathing assessed by Nijmegen breathing questionnaire at week 4 and week 12 | baseline, week 4, week 12
  the total score ranges from 0 to 64 points with higher scores indicating hyperventilation
Change from baseline chronic fatigue syndrome assessed by fatigue assessment scale at week 4 and week 12 | baseline, week 4, week 12
  the total score ranges from 10 to 50 points with higher scores indicating more fatigue
Change from baseline chronic fatigue syndrome assessed by canadian consensus criteria at week 12 | baseline, week 12
  the canadian consensus criteria indicate if patients developed a chronic fatigue syndrome/myalgic encephalomyelitis
Change from baseline functional status assessed by post-COVID functional status scale at week 4 and week 12 | baseline, week 4, week 12
  the total score ranges from 0 to 4 points with higher scores indicating more impairment
Change from baseline physical activity assessed by Garmin watch at week 4 and week 12 | baseline, week 4, week 12
  daily total steps per day will be recorded by a Garmin watch linked to the SaniQ App
Change from baseline blood pressure assessed at week 4 and week 12 | baseline, week 4, week 12
  blood pressure will be measured at the upper arm using the Aponorm device
Change from baseline oxygen saturation assessed by pulse oximeter at week 4 and week 12 | baseline, week 4, week 12
  Beurer pulse oximeter
Change from baseline peak flow assessed by peak flow meter at week 4 and week 12 | baseline, week 4, week 12
  peak flow will be assessed by smart one spirometer

CONTACTS AND LOCATIONS:
Locations (8):
- Germany (8):
  - University Hospital Augsburg, Augsburg
  - Praxis Dr. Schrag, Bad Reichenhall
  - Pneumologen Lichterfelde Berlin, Berlin
  - Praxis im Zentrum Erlangen, Erlangen
  - Pneumopraxis Marburg, Marburg
  - Lungenärzte am Rundfunkplatz, München, Munich
  - COVID ambulance Prof. Koczulla, Schönau am Königssee
  - Praxis Dr. Roch, Schwabach

IPD SHARING:
Plan to Share IPD: Undecided